CLINICAL TRIAL: NCT03662334
Title: A Phase 4, Double Blind, Single Center, Randomized, Cross-Over Study of Continuous Subcutaneous Insulin Infusion (CSII) Pump Functionality in Subjects With Type 1 Diabetes Comparing Pretreatment vs. No Pretreatment With Recombinant Human Hyaluronidase (rHuPH20)
Brief Title: A Study of Continuous Subcutaneous Insulin Infusion (CSII) Pump Function in Subjects With Type 1 Diabetes With Recombinant Human Hyaluronidase (rHuPH20)
Acronym: HALO-117-406
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HALO-117-406
Record Dates: First submitted 2018-08-13; First posted 2018-09-07 (Actual); Results first posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes; Type 1 Diabetes Mellitus; Type 1 Diabetes; T1DM; Continuous Subcutaneous Insulin Infusion (CSII); CSII; Insulin pump; Insulin; rHuPH20; Hylenex; recombinant human hyaluronidase (rHuPH20); Recombinant hyaluronidase
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance | interventions — Insulin, Short-Acting; Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hylenex recombinant (Experimental): Comparing the preadministration of Hylenex recombinant in the setting of continuous subcutaneous insulin infusion (CSII).
  Interventions: Drug: Rapid Acting insulin with pre-treatment of rHuPH20
- Sham Injection (Sham Comparator): Comparing the preadministration of a sham injection in the setting of CSII.
  Interventions: Device: Sham injection

INTERVENTIONS:
Drug: Rapid Acting insulin with pre-treatment of rHuPH20 — Hylenex recombinant will be administered via infusion sets and insulin pumps. These will be compatible with component tubing system attached to the insulin infusion site and will be placed in the lower abdominal area.
  Other Names: Humalog; Hylenex
  Arms: Hylenex recombinant
Device: Sham injection — A sham injection will be administered via infusion sets and insulin pumps. These will be compatible with component tubing system attached to the insulin infusion site and will be placed in the lower abdominal area.
  Other Names: placebo
  Arms: Sham Injection

SUMMARY:
The goal of this study is to determine if Hylenex recombinant leads to changes in the insulin time-action profiles and glucose responses when preadministered in the setting of continuous subcutaneous insulin infusion (CSII) compared to CSII without Hylenex recombinant (sham injection).

DETAILED DESCRIPTION:
There is a recognized need for more rapid insulin action than is available from current rapid-acting analog products. In addition, current products have inconstant absorption and action profiles over the course of infusion set life. Previous human studies of prandial insulin preparations have used co-mixtures of rHuPH20 (study drug) with insulin delivered to study participants by subcutaneous injection and have demonstrated acceleration of insulin absorption and action. CSII has been used clinically for the treatment of diabetes over the last three decades, and a previous study using a co-mixture of rHuPH20 during CSII showed that the combination resulted in a more consistent and ultrafast profile of insulin absorption and action across infusion set use as compared to rapid analog insulin alone.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants between the ages 18 and 65 years, inclusive.
2. Females of child-bearing potential must agree to use a standard and effective means of birth control for the duration of the study. Adequate contraceptive measures include oral or injectable contraceptives, sterilization, intra-uterine device (IUD), barrier methods, or abstinence.
3. Participants with type 1 diabetes mellitus treated with insulin (multiple daily injections or continuous subcutaneous insulin infusion [CSII]) diagnosed ≥ 12 months prior to enrollment
4. Body mass index (BMI) 18.0 to 32.0 kilograms per meters squared (kg/m^2)
5. HbA1c (glycated hemoglobin A1c) ≤ 10% based on local laboratory results
6. Fasting C-peptide < 0.6 nanograms per milliliter (ng/mL)
7. Current treatment with insulin <1.2 Units per kg per day (U/kg/day)
8. Participant should be in good general health based on medical history and physical examination, without medical conditions that might prevent the completion of study drug injections and assessments required in this protocol

Exclusion Criteria:

1. Inability to comply with study requirements as judged by the Investigator
2. Known or suspected allergy to any component of any of the study drugs in this trial
3. A participant who has proliferative retinopathy or maculopathy, severe gastroparesis, and/or severe neuropathy, in particular autonomic neuropathy, as judged by the Investigator
4. As judged by the Investigator, clinically significant active disease of the gastrointestinal, cardiovascular (including a history of arrhythmia or conduction delays on electrocardiogram), hepatic, neurological, renal, genitourinary, or hematological systems
5. As judged by the Investigator, uncontrolled hypertension (diastolic blood pressure ≥ 100 millimeters of mercury [mmHg] and/or systolic blood pressure ≥ 160 mmHg after 5 minutes in the supine position)
6. History of any illness or disease that in the opinion of the Investigator might confound the results of the trial or pose additional risk in administering the study drugs to the participant
7. As judged by the Investigator, clinically significant findings in routine laboratory data. Anemia with hemoglobin less than lower limits of normal at screening is specifically exclusionary
8. Use of drugs that may interfere with the interpretation of trial results or are known to cause clinically relevant interference with insulin action, glucose utilization, or recovery from hypoglycemia, or drugs not permitted according to Hylenex recombinant package insert
9. Recurrent major hypoglycemia or hypoglycemic unawareness, as judged by the Investigator
10. Current addiction to alcohol or substances of abuse as determined by the Investigator
11. Blood donation (> 500 mL) within the previous 8 weeks (56 days) prior to Day -1 of Treatment Period 1
12. Pregnancy, breast-feeding, the intention of becoming pregnant, or not using adequate contraceptive measures (adequate contraceptive measures consist of sterilization, IUD, oral or injectable contraceptives, or barrier methods)
13. Mental incapacity, unwillingness, or language barriers precluding adequate understanding or cooperation in this study
14. Participation in any other clinical trial and receipt of any investigational drug within 4 weeks of Day -1 of Treatment Period 1
15. Any condition (intrinsic or extrinsic) that in the judgment of the Investigator will interfere with trial participation or evaluation of data
16. Positive for human immunodeficiency virus (HIV), Hepatitis C or Hepatitis B
17. Tobacco and nicotine use within 3 months prior to Day 1 of Treatment Period 1 or use during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-10-03 (Actual); Primary Completion 2014-02-27 (Actual); Study Completion 2014-02-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Profil Institute for Clinical Research, Chula Vista, California, United States

REFERENCES:
- See also: Halozyme Therapeutics — http://www.halozyme.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All three parts (Parts 1, 2, and 3) of this exploratory study were to use a cross-over design that would maximize efficiency while minimizing sample size. Only Part 2 of this study was conducted; thus, all 14 participants were enrolled in Part 2 only.
Groups:
- Hyaluronidase Human Injection/Sham Injection: Participants received pretreatment of 1 milliliter (mL) hyaluronidase human injection on Day 1 of Treatment Period 1. After a 3- to 7-day washout period, participants received pretreatment of 1 mL sham injection on Day 1 of Treatment Period 2.
- Sham Injection/Hyaluronidase Human Injection: Participants received pretreatment of 1 mL sham injection on Day 1 of Treatment Period 1. After a 3- to 7-day washout period, participants received pretreatment of 1 mL hyaluronidase human injection on Day 1 of Treatment Period 2.
Period: Part 1: Treatment Period 1
Arm/Group | Hyaluronidase Human Injection/Sham Injection | Sham Injection/Hyaluronidase Human Injection
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0
Period: Part 1: Treatment Period 2
Arm/Group | Hyaluronidase Human Injection/Sham Injection | Sham Injection/Hyaluronidase Human Injection
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0
Period: Part 2: Treatment Period 1 (2 Days)
Arm/Group | Hyaluronidase Human Injection/Sham Injection | Sham Injection/Hyaluronidase Human Injection
Started | 7 (Part 1 of the study was not conducted. Participants were enrolled starting with Part 2.) | 7 (Part 1 of the study was not conducted. Participants were enrolled starting with Part 2.)
Completed | 7 | 7
Not Completed | 0 | 0
Period: Part 2: Treatment Period 2 (2 Days)
Arm/Group | Hyaluronidase Human Injection/Sham Injection | Sham Injection/Hyaluronidase Human Injection
Started | 7 | 7
Completed | 6 | 7
Not Completed | 1 | 0
Not completed — Intended Changes to Clamp Procedure | 1 | 0
Period: Part 3: Treatment Period 1
Arm/Group | Hyaluronidase Human Injection/Sham Injection | Sham Injection/Hyaluronidase Human Injection
Started | 0 (Part 3 of the study was not conducted. No participants were enrolled in this part of the study.) | 0 (Part 3 of the study was not conducted. No participants were enrolled in this part of the study.)
Completed | 0 | 0
Not Completed | 0 | 0
Period: Part 3: Treatment Period 2
Arm/Group | Hyaluronidase Human Injection/Sham Injection | Sham Injection/Hyaluronidase Human Injection
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data were collected in members of the Safety Population, comprised of all randomized participants exposed to at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hyaluronidase Human Injection/Sham Injection | Sham Injection/Hyaluronidase Human Injection | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (8.90) | 40.4 (14.84) | 42.0 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 5 | 5 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Area Under the Curve (AUC) of Glucose Infusion Rate (GIR) From 0-6 Hours
Time Frame: 0-6 hours
Population: The study was stopped early, prior to enrolling the planned 24 participants. As a result, data were not collected for analysis of this outcome measure. Only Part 2 of the study was conducted.
Arm/Group | Hyaluronidase Human Injection/Sham Injection | Sham Injection/Hyaluronidase Human Injection
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Part 2: Time to Reduction in Plasma Glucose by 80 Milligrams Per Deciliter (mg/dL) Following CSII Bolus
Description: Time to reduction is reported as the maximum time it took for any participant receiving each treatment sequence to achieve a reduction in plasma glucose by 80 mg/dL. During the course of the study, it became difficult to establish a stable hyperglycemic plateau with a target glucose level of 220 mg/dL, even after adjusting several operational parameters. The study was stopped early, prior to enrolling the planned 24 participants for Part 2. Thus, analysis for this endpoint was not conducted. Raw data (as a maximum) are reported.
Time Frame: 0-10 hours
Population: Safety Population: all randomized participants exposed to at least one dose of study drug
Measure: Number; unit: hours
Arm/Group | Hyaluronidase Human Injection/Sham Injection | Sham Injection/Hyaluronidase Human Injection
Number analyzed (Participants) | 7 | 7
hours
  First Intervention | 5.58 | 5.23
  Second Intervention | 4.63 | 5.32

3. Primary Outcome: Part 3: Time to Achieve Plasma Glucose >90 mg/dL After Release of Hypoglycemic CSII Clamp
Time Frame: 0-12 hours
Population: as for outcome 1
Arm/Group | Hyaluronidase Human Injection/Sham Injection | Sham Injection/Hyaluronidase Human Injection
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Part 1: Time-action Profile, Assessed by GIR in Euglycemic Participants
Time Frame: up to approximately 10 hours
Population: as for outcome 1
Arm/Group | Hyaluronidase Human Injection/Sham Injection | Sham Injection/Hyaluronidase Human Injection
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Part 1: Mean Maximum Concentration (Cmax)
Time Frame: up to approximately 22 hours
Population: as for outcome 1
Arm/Group | Hyaluronidase Human Injection/Sham Injection | Sham Injection/Hyaluronidase Human Injection
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Part 1: Time to Achieve Maximum Concentration (Tmax)
Time Frame: up to approximately 22 hours
Population: as for outcome 1
Arm/Group | Hyaluronidase Human Injection/Sham Injection | Sham Injection/Hyaluronidase Human Injection
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Part 1: Early Time to 50% Maximum Serum Insulin Concentration (t50%) Max
Time Frame: up to approximately 22 hours
Population: as for outcome 1
Arm/Group | Hyaluronidase Human Injection/Sham Injection | Sham Injection/Hyaluronidase Human Injection
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Part 1: Time to 50% of Total AUC (AUC0-last)
Time Frame: up to approximately 22 hours
Population: as for outcome 1
Arm/Group | Hyaluronidase Human Injection/Sham Injection | Sham Injection/Hyaluronidase Human Injection
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Part 1: Fractional and Absolute AUC0-1hr
Time Frame: 0 to 1 hour
Population: as for outcome 1
Arm/Group | Hyaluronidase Human Injection/Sham Injection | Sham Injection/Hyaluronidase Human Injection
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Part 1: Fractional and Absolute AUC2hr-end
Time Frame: 2 to approximately 22 hours
Population: as for outcome 1
Arm/Group | Hyaluronidase Human Injection/Sham Injection | Sham Injection/Hyaluronidase Human Injection
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Part 1: Area Under the Curve From Time Zero to the Last Measureable Concentration (AUC0-last)
Time Frame: up to approximately 22 hours
Population: as for outcome 1
Arm/Group | Hyaluronidase Human Injection/Sham Injection | Sham Injection/Hyaluronidase Human Injection
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Part 1: Mean Residence Time (MRT)
Time Frame: up to approximately 22 hours
Population: as for outcome 1
Arm/Group | Hyaluronidase Human Injection/Sham Injection | Sham Injection/Hyaluronidase Human Injection
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Part 2: Plasma Glucose Concentration Over Time
Description: Plasma glucose concentration over time is reported as the maximum concentration for any participant receiving each treatment sequence. During the course of the study, it became difficult to establish a stable hyperglycemic plateau with a target glucose level of 220 mg/dL, even after adjusting several operational parameters. The study was stopped early, prior to enrolling the planned 24 participants for Part 2. Thus, analysis for this endpoint was not conducted. Raw data (as a maximum) are reported.
Time Frame: up to approximately 10 hours
Population: Safety Population
Measure: Number; unit: mg/dL
Arm/Group | Hyaluronidase Human Injection/Sham Injection | Sham Injection/Hyaluronidase Human Injection
Number analyzed (Participants) | 7 | 7
mg/dL
  First Intervention | 299 | 341
  Second Intervention | 350 | 445

14. Secondary Outcome: Part 2: Insulin Analog Serum Concentration as a Function of Time Following Bolus Insulin Infusion
Description: Insulin analog serum concentration is reported as the maximum concentration for any participant receiving each treatment sequence. During the course of the study, it became difficult to establish a stable hyperglycemic plateau with a target glucose level of 220 mg/dL, even after adjusting several operational parameters. The study was stopped early, prior to enrolling the planned 24 participants for Part 2. Thus, analysis for this endpoint was not conducted. Raw data (as a maximum) are reported.
Time Frame: up to approximately 10 hours
Population: Safety Population
Measure: Number; unit: picomolar
Arm/Group | Hyaluronidase Human Injection/Sham Injection | Sham Injection/Hyaluronidase Human Injection
Number analyzed (Participants) | 7 | 7
picomolar
  First Intervention | 1341.8 | 805.1
  Second Intervention | 688.5 | 1092.6

15. Secondary Outcome: Part 3: Plasma Glucose Concentration Over Time
Time Frame: up to approximately 12 hours
Population: as for outcome 1
Arm/Group | Hyaluronidase Human Injection/Sham Injection | Sham Injection/Hyaluronidase Human Injection
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Part 3: Insulin Analog Serum Concentration as a Function of Time Following Termination of Insulin Infusion
Time Frame: up to approximately 12 hours
Population: as for outcome 1
Arm/Group | Hyaluronidase Human Injection/Sham Injection | Sham Injection/Hyaluronidase Human Injection
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 155 days
Groups:
- Hyaluronidase Human Injection: Participants received pretreatment of 1 milliliter (mL) hyaluronidase human injection on Day 1 of either Treatment Period 1 or Treatment Period 2. The two periods were separated by a 3- to 7-day washout period.
- Sham Injection: Participants received pretreatment of 1 mL sham injection on Day 1 of either Treatment Period 1 or Treatment Period 2. The two periods were separated by a 3- to 7-day washout period.
Arm/Group | Hyaluronidase Human Injection | Sham Injection
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 4/14 | 2/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hyaluronidase Human Injection (N=14) | Sham Injection (N=14)
Injection Site Pain (General disorders) | 2 | 0
Injection Site Haematoma (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
During the course of the study, it became difficult to establish a stable hyperglycemic plateau with a target glucose level of 220 milligrams per deciliter. The study was stopped early, prior to enrolling the planned 24 participants for Part 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information obtained as a result of this study or during the conduct of this study will be regarded as confidential. The Investigator agrees to use the information for the purpose of carrying out this study and for no other purpose, unless written permission from the sponsor (Halozyme) is obtained.